CLINICAL TRIAL: NCT06344234
Title: Noninvasive Assessment of Inspiratory Effort and Tidal Distension During Noninvasive Ventilation. The INSPIRE Study.
Brief Title: Non-invasive Assessment of Inspiratory Effort and Tidal Distension During Non-invasive Ventilation (INSPIRE)
Acronym: INSPIRE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, Professor, University of Bari
Other Study IDs: 0049191
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Disease; Artificial Respiration
Keywords: noninvasive ventilation; respiration, artificial; Ventilators, Mechanical; Positive End-Expiratory Pressure
MeSH Terms: conditions — Respiration Disorders; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort (n=60): All hypoxemic patients with a PaO2/FiO2 ratio equal or lower than 300, receiving post-extubation noninvasive ventilation.
  Participants will undergo the following tasks and treatments:
  * Complete written informed consent before enrollment.
  * Post-extubation noninvasive ventilation via nose-to-mouth and full-face masks.
  * Monitoring of esophageal pressure
  * Continuous recording of airway pressure, flow, and esophageal pressure (Pes), using a dedicated pneumotachograph and pressure transducer.
  * Sudden end-inspiratory and end-expiratory occlusion maneuvers.
  * Collection of hemodynamic and arterial blood-gas parameters, performed according to clinical judgment, along with assessments of dyspnea and discomfort using a modified visual analogue scale (VAS).
  * Diaphragm ultrasound during occlusion maneuvers, measuring diaphragm displacement, diaphragm thickening fraction (DTF%), and diaphragmatic excursion (Ex) under various conditions.
  Interventions: Diagnostic Test: End-inspiratory Maneuvers

INTERVENTIONS:
Diagnostic Test: End-inspiratory Maneuvers — Airway pressure, flow, and esophageal pressure will be continuously recorded in all patients using a dedicated pneumotachograph and pressure transducer: all signals will be acquired and stored. Once a stable ventilation pattern is observed NIV will be administered by setting ventilator in invasive-pressure support ventilation. PEEP and PS-level will by kept constant while expiratory trigger will be adjusted to optimize patient-ventilatory synchrony. Immediately after, sudden end-inspiratory and end-expiratory occlusion maneuvers will be performed to measure plateau pressure and end-expiratory airway occlusion pressure (ΔPocc), respectively. Invasive PSV will be used only to perform the occlusion maneuvers, subsequently, PSV will be delivered in non-invasive PSV mode. Patient's blood-gas parameters and vital signs will be collected, including discomfort assessment. During the occlusion maneuvers, diaphragm ultrasound will be performed, and images will be recorded.
  Other Names: End-Expiratory Occlusion Maneuvers; Esophageal pressure monitoring; Diaphragmatic ultrasounds

SUMMARY:
The goal of this observational study is to evaluate whether the airway occlusion pressure recorded during a sudden end-expiratory breath-hold (ΔPocc) is correlated with esophageal swing in pressure and the reliability of P0.1, driving pressure, plateau pressure, pressure-muscle index, and diaphragm ultrasound as noninvasive estimates of inspiratory effort and lung distension in hypoxemic patients undergoing NIV.

The main questions this trial aims to answer are:

- Primary Outcome: whether the airway occlusion pressure recorded during a sudden end-expiratory breath-hold (ΔPocc) is correlated with esophageal swing in pressure and the reliability of various noninvasive estimates of inspiratory effort and lung distension in hypoxemic patients undergoing NIV.

Secondary outcomes will include:

* Statistic metric of association between P0.1, ΔP, PMI and ΔPes
* Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and PaO2/FiO2 ratio
* Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and tidal volume
* Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and DTF%
* Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and Ex/DTF%
* Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and respiratory rate, VAS dyspnea and VAS discomfort.

Participants will undergo the following tasks and treatments:

* Complete written informed consent before enrollment.
* Post-extubation noninvasive ventilation via nose-to-mouth and full-face masks.
* Monitoring of esophageal pressure (in all patients the catheter will be placed before extubation, according to clinical judgment, and its correct position will be verified through a positive pressure occlusion test)
* Continuous recording of airway pressure, flow, and esophageal pressure (Pes), using a dedicated pneumotachograph and pressure transducer.
* Sudden end-inspiratory and end-expiratory occlusion maneuvers, to measure plateau pressure (Pplat) and end-expiratory airway occlusion pressure (ΔPocc), respectively.
* Collection of hemodynamic and arterial blood-gas parameters, performed according to clinical judgment, along with assessments of dyspnea and discomfort using a modified visual analogue scale (VAS).
* Diaphragm ultrasound during occlusion maneuvers, measuring diaphragm displacement, diaphragm thickening fraction (DTF%), and diaphragmatic excursion (Ex) under various conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Non-pregnant and non-lactating.
* Monitored through esophageal pressure for clinical decision before extubation.
* Able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients with severe facial trauma or deformity that precludes the placement of a facemask or esophageal catheter.
* Patients with neuromuscular disorders that may impair inspiratory drive and effort.
* Patients with acute exacerbation of COPD
* Patients with esophageal or tracheal abnormalities that impede esophageal manometry.
* Patients with a known hypersensitivity or allergy to any of the materials used in the study.
* Excessive air leak (difference between inspiratory and expiratory tidal volume major or equal to 30% [prot. n 1136947]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All hypoxemic patients with a PaO2/FiO2 ratio equal or lower than 300, receiving post-extubation noninvasive ventilation via an nose-to-mouth or a full-face mask, will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Statistic metric of association between ΔPocc and ΔPes | 24 hours
  to evaluate whether the airway occlusion pressure recorded during a sudden end-expiratory breath-hold (ΔPocc) is correlated with esophageal swing in pressure

SECONDARY OUTCOMES:
Statistic metric of association between P0.1, ΔP, PMI and ΔPes | 24 hours
Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and PaO2/FiO2 ratio | 24 hours
Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and tidal volume | 24 hours
Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and DTF% | 24 hours
Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and Ex/DTF% | 24 hours
Statistic metric of association between P0.1, ΔPocc, ΔP, PMI and respiratory rate, VAS dyspnea and VAS discomfort | 24 hours

OTHER OUTCOMES:
Reliability of various noninvasive estimates of inspiratory effort and lung distension in hypoxemic patients undergoing NIV | 24 hours
  To investigate the reliability of P0.1, driving pressure, plateau pressure, pressure-muscle index, and diaphragm ultrasound as noninvasive estimates of inspiratory effort and lung distension in hypoxemic patients undergoing NIV

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grasso, Prof, Study Chair — Azienda Ospedaliero-Universitaria "Consorziale Policlinico" Bari
Locations (1):
- Azienda ospedaliero-universitaria consorziale policlinico di Bari, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grieco DL, Menga LS, Cesarano M, Rosa T, Spadaro S, Bitondo MM, Montomoli J, Falo G, Tonetti T, Cutuli SL, Pintaudi G, Tanzarella ES, Piervincenzi E, Bongiovanni F, Dell'Anna AM, Delle Cese L, Berardi C, Carelli S, Bocci MG, Montini L, Bello G, Natalini D, De Pascale G, Velardo M, Volta CA, Ranieri VM, Conti G, Maggiore SM, Antonelli M; COVID-ICU Gemelli Study Group. Effect of Helmet Noninvasive Ventilation vs High-Flow Nasal Oxygen on Days Free of Respiratory Support in Patients With COVID-19 and Moderate to Severe Hypoxemic Respiratory Failure: The HENIVOT Randomized Clinical Trial. JAMA. 2021 May 4;325(17):1731-1743. doi: 10.1001/jama.2021.4682. PMID 33764378
- [Background] Grasselli G, Calfee CS, Camporota L, Poole D, Amato MBP, Antonelli M, Arabi YM, Baroncelli F, Beitler JR, Bellani G, Bellingan G, Blackwood B, Bos LDJ, Brochard L, Brodie D, Burns KEA, Combes A, D'Arrigo S, De Backer D, Demoule A, Einav S, Fan E, Ferguson ND, Frat JP, Gattinoni L, Guerin C, Herridge MS, Hodgson C, Hough CL, Jaber S, Juffermans NP, Karagiannidis C, Kesecioglu J, Kwizera A, Laffey JG, Mancebo J, Matthay MA, McAuley DF, Mercat A, Meyer NJ, Moss M, Munshi L, Myatra SN, Ng Gong M, Papazian L, Patel BK, Pellegrini M, Perner A, Pesenti A, Piquilloud L, Qiu H, Ranieri MV, Riviello E, Slutsky AS, Stapleton RD, Summers C, Thompson TB, Valente Barbas CS, Villar J, Ware LB, Weiss B, Zampieri FG, Azoulay E, Cecconi M; European Society of Intensive Care Medicine Taskforce on ARDS. ESICM guidelines on acute respiratory distress syndrome: definition, phenotyping and respiratory support strategies. Intensive Care Med. 2023 Jul;49(7):727-759. doi: 10.1007/s00134-023-07050-7. Epub 2023 Jun 16. PMID 37326646
- [Background] Bellani G, Laffey JG, Pham T, Madotto F, Fan E, Brochard L, Esteban A, Gattinoni L, Bumbasirevic V, Piquilloud L, van Haren F, Larsson A, McAuley DF, Bauer PR, Arabi YM, Ranieri M, Antonelli M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Noninvasive Ventilation of Patients with Acute Respiratory Distress Syndrome. Insights from the LUNG SAFE Study. Am J Respir Crit Care Med. 2017 Jan 1;195(1):67-77. doi: 10.1164/rccm.201606-1306OC. PMID 27753501
- [Background] Menga LS, Cese LD, Bongiovanni F, Lombardi G, Michi T, Luciani F, Cicetti M, Timpano J, Ferrante MC, Cesarano M, Anzellotti GM, Rosa T, Natalini D, Tanzarella ES, Cutuli SL, Pintaudi G, De Pascale G, Dell'Anna AM, Bello G, Pennisi MA, Maggiore SM, Maviglia R, Grieco DL, Antonelli M. High Failure Rate of Noninvasive Oxygenation Strategies in Critically Ill Subjects With Acute Hypoxemic Respiratory Failure Due to COVID-19. Respir Care. 2021 May;66(5):705-714. doi: 10.4187/respcare.08622. Epub 2021 Mar 2. PMID 33653913
- [Background] Grieco DL, Menga LS, Eleuteri D, Antonelli M. Patient self-inflicted lung injury: implications for acute hypoxemic respiratory failure and ARDS patients on non-invasive support. Minerva Anestesiol. 2019 Sep;85(9):1014-1023. doi: 10.23736/S0375-9393.19.13418-9. Epub 2019 Mar 12. PMID 30871304
- [Background] Chi Y, Zhao Z, Frerichs I, Long Y, He H. Prevalence and prognosis of respiratory pendelluft phenomenon in mechanically ventilated ICU patients with acute respiratory failure: a retrospective cohort study. Ann Intensive Care. 2022 Mar 5;12(1):22. doi: 10.1186/s13613-022-00995-w. PMID 35246748
- [Background] Goligher EC, Jonkman AH, Dianti J, Vaporidi K, Beitler JR, Patel BK, Yoshida T, Jaber S, Dres M, Mauri T, Bellani G, Demoule A, Brochard L, Heunks L. Clinical strategies for implementing lung and diaphragm-protective ventilation: avoiding insufficient and excessive effort. Intensive Care Med. 2020 Dec;46(12):2314-2326. doi: 10.1007/s00134-020-06288-9. Epub 2020 Nov 2. PMID 33140181
- [Background] Spinelli E, Mauri T, Beitler JR, Pesenti A, Brodie D. Respiratory drive in the acute respiratory distress syndrome: pathophysiology, monitoring, and therapeutic interventions. Intensive Care Med. 2020 Apr;46(4):606-618. doi: 10.1007/s00134-020-05942-6. Epub 2020 Feb 3. PMID 32016537
- [Background] Tonelli R, Fantini R, Tabbi L, Castaniere I, Pisani L, Pellegrino MR, Della Casa G, D'Amico R, Girardis M, Nava S, Clini EM, Marchioni A. Early Inspiratory Effort Assessment by Esophageal Manometry Predicts Noninvasive Ventilation Outcome in De Novo Respiratory Failure. A Pilot Study. Am J Respir Crit Care Med. 2020 Aug 15;202(4):558-567. doi: 10.1164/rccm.201912-2512OC. PMID 32325004
- [Background] Menga LS, Delle Cese L, Rosa T, Cesarano M, Scarascia R, Michi T, Biasucci DG, Ruggiero E, Dell'Anna AM, Cutuli SL, Tanzarella ES, Pintaudi G, De Pascale G, Sandroni C, Maggiore SM, Grieco DL, Antonelli M. Respective Effects of Helmet Pressure Support, Continuous Positive Airway Pressure, and Nasal High-Flow in Hypoxemic Respiratory Failure: A Randomized Crossover Clinical Trial. Am J Respir Crit Care Med. 2023 May 15;207(10):1310-1323. doi: 10.1164/rccm.202204-0629OC. PMID 36378814
- [Background] Yoshida T, Grieco DL, Brochard L, Fujino Y. Patient self-inflicted lung injury and positive end-expiratory pressure for safe spontaneous breathing. Curr Opin Crit Care. 2020 Feb;26(1):59-65. doi: 10.1097/MCC.0000000000000691. PMID 31815775
- [Background] Bertoni M, Spadaro S, Goligher EC. Monitoring Patient Respiratory Effort During Mechanical Ventilation: Lung and Diaphragm-Protective Ventilation. Crit Care. 2020 Mar 24;24(1):106. doi: 10.1186/s13054-020-2777-y. PMID 32204729
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Background] Mojoli F, Torriglia F, Orlando A, Bianchi I, Arisi E, Pozzi M. Technical aspects of bedside respiratory monitoring of transpulmonary pressure. Ann Transl Med. 2018 Oct;6(19):377. doi: 10.21037/atm.2018.08.37. PMID 30460251
- [Background] Dianti J, Bertoni M, Goligher EC. Monitoring patient-ventilator interaction by an end-expiratory occlusion maneuver. Intensive Care Med. 2020 Dec;46(12):2338-2341. doi: 10.1007/s00134-020-06167-3. Epub 2020 Jul 4. No abstract available. PMID 32623476
- [Background] Whitelaw WA, Derenne JP, Milic-Emili J. Occlusion pressure as a measure of respiratory center output in conscious man. Respir Physiol. 1975 Mar;23(2):181-99. doi: 10.1016/0034-5687(75)90059-6. PMID 1144940
- [Background] Telias I, Damiani F, Brochard L. The airway occlusion pressure (P0.1) to monitor respiratory drive during mechanical ventilation: increasing awareness of a not-so-new problem. Intensive Care Med. 2018 Sep;44(9):1532-1535. doi: 10.1007/s00134-018-5045-8. Epub 2018 Jan 19. No abstract available. PMID 29350241
- [Background] Bellani G, Grassi A, Sosio S, Foti G. Plateau and driving pressure in the presence of spontaneous breathing. Intensive Care Med. 2019 Jan;45(1):97-98. doi: 10.1007/s00134-018-5311-9. Epub 2018 Jul 13. No abstract available. PMID 30006893
- [Background] Foti G, Cereda M, Banfi G, Pelosi P, Fumagalli R, Pesenti A. End-inspiratory airway occlusion: a method to assess the pressure developed by inspiratory muscles in patients with acute lung injury undergoing pressure support. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 1):1210-6. doi: 10.1164/ajrccm.156.4.96-02031. PMID 9351624
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Dube BP, Dres M, Mayaux J, Demiri S, Similowski T, Demoule A. Ultrasound evaluation of diaphragm function in mechanically ventilated patients: comparison to phrenic stimulation and prognostic implications. Thorax. 2017 Sep;72(9):811-818. doi: 10.1136/thoraxjnl-2016-209459. Epub 2017 Mar 30. PMID 28360224
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Chiumello D, Consonni D, Coppola S, Froio S, Crimella F, Colombo A. The occlusion tests and end-expiratory esophageal pressure: measurements and comparison in controlled and assisted ventilation. Ann Intensive Care. 2016 Dec;6(1):13. doi: 10.1186/s13613-016-0112-1. Epub 2016 Feb 12. PMID 26868503